CLINICAL TRIAL: NCT07280962
Title: Comparison of Outcomes Between Packing Versus no Packing in Perianal Abscess Cavity After Incision and Drainage
Brief Title: Packing Versus no Packing in Perianal Abscess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr. Hafsa Khan
Record Dates: First submitted 2025-11-23; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Perianal Abccess
Keywords: Perianal abccess

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Packing group (Active Comparator): This group will undergo packing of perianal abccess after the drainage.
  Interventions: Procedure: Packing of perianal abccess with surgical gauze
- Non-packing group (Placebo Comparator): This group received no packing after drainage of perianal abcess.
  Interventions: Procedure: Non-packing of perianal abccess

INTERVENTIONS:
Procedure: Packing of perianal abccess with surgical gauze — Patients will undergo packing of perianal abcess after incision and drainage
  Arms: Packing group
Procedure: Non-packing of perianal abccess — The patients in non-packing group received no packing of wound after drainage of parianal abccess.
  Arms: Non-packing group

SUMMARY:
Perianal abscess is a common surgical emergency that causes significant pain and discomfort. The standard treatment involves incision and drainage (I&D) of the abscess cavity, traditionally followed by packing to prevent re-accumulation of pus and to promote healing. However, packing is often painful, requires frequent dressing changes, and increases patient discomfort as well as healthcare costs. Recent studies suggest that leaving the cavity unpacked may result in similar healing outcomes while reducing postoperative pain and shortening the length of hospital stay. This randomized controlled trial aims to compare the outcomes of packing versus no packing of the perianal abscess cavity following I&D. The study will evaluate postoperative pain using the Visual Analogue Scale at 6, 12, and 24 hours, duration of hospital stay, and the recurrence rate within one month. The findings of this research are expected to guide evidence-based clinical practice by improving patient comfort, reducing hospital burden, and optimizing postoperative care protocols.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to evaluate and compare the clinical outcomes of packing versus no packing of the perianal abscess cavity following incision and drainage (I&D), the standard surgical management for this common anorectal condition. Perianal abscesses develop due to infection and obstruction of the anal glands, resulting in severe pain, swelling, and systemic discomfort. Traditionally, postoperative packing of the abscess cavity has been performed to maintain drainage, achieve hemostasis, and prevent re-accumulation of pus; however, this practice is associated with considerable pain, delayed wound healing, repeated dressing changes, and increased hospital visits. In contrast, leaving the cavity unpacked and allowing healing by secondary intention may minimize patient discomfort, reduce healthcare costs, and shorten recovery time without increasing the risk of recurrence.

This study will be conducted among adult patients diagnosed with perianal abscess requiring I&D, who will be randomly assigned to two groups: Group A (packing) and Group B (no packing). Postoperative pain will be assessed using the Visual Analogue Scale (VAS) at 6, 12, and 24 hours after the procedure. The duration of hospital stay and recurrence of the abscess within one month will also be recorded. Data will be analyzed using SPSS software, applying independent t-tests and chi-square tests to determine statistical significance, with a p-value < 0.05 considered significant. The findings of this study are expected to provide evidence-based insights into whether non-packing offers comparable or superior outcomes to conventional packing, ultimately guiding surgical practice toward safer, more comfortable, and cost-effective patient care.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting in the emergency department diagnosed with acute perianal abscess (Diagnosed on the basis of history and clinical examination with ultrasonographic evidence of quantifiable collection and confirmed by needle aspiration of pus from swelling) based on history and examination, requiring incision and drainage.

Exclusion Criteria:

* Patients with prior perianal fistulas based on history and examination
* Patients with recurrent abscess (based on history)
* Horseshoe abscess as based on examination
* Previous pelvic irradiation (based on history)
* Immunocompromised patients
* Malignant abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Post-operative Pain | 24 hours
  Patients was assessed for the post-operative pain by using VAS. VAS is a tool used to assess the intensity of pain in patients. The scoring ranges from 0-10, where 0 is minimum or no pain and 10 is maximum pain.

SECONDARY OUTCOMES:
Recurrence | 1 month
  Recurrence will be labeled in a patient at 1 month follow-up period after incision and drainage if the patient complains of pain and fever, induration, and tenderness at the operated site, labeled as a perianal abscess at the same site, requiring incision and drainage.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perera AP, Howell AM, Sodergren MH, Farne H, Darzi A, Purkayastha S, Paraskeva P. A pilot randomised controlled trial evaluating postoperative packing of the perianal abscess. Langenbecks Arch Surg. 2015 Feb;400(2):267-71. doi: 10.1007/s00423-014-1231-5. Epub 2014 Jul 23. PMID 25053508
- See also: This study elaborates the outcomes of role of packing in perianal abcess. — https://pmc.ncbi.nlm.nih.gov/articles/PMC10364677
- Available data/document: Study Protocol — https://heyzine.com/flip-book/0d5ec370d6.html — https://heyzine.com/flip-book/0d5ec370d6.html